CLINICAL TRIAL: NCT00126867
Title: Thymidylate Synthase Polymorphisms as a Predictor of Toxicity to Capecitabine Based Adjuvant Chemotherapy in Colon Cancer Treatment
Brief Title: Thymidylate Synthase Polymorphisms as a Predictor of Toxicity to Capecitabine Chemotherapy in Colon Cancer Treatment
Status: Terminated | Type: Observational
Why Stopped: Insufficient accrual and no funding
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: GI-05-0049 / 21882
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Colon Cancer
Keywords: thymidylate synthase polymers; rapecitabine; adjuvant; colon cancer; toxicity; Stage II colon cancer; Stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cancers of the colon and rectum are the third most common cancers in Canadian males and females. The initial therapy of colorectal cancer is surgery to remove the cancer and nearby lymph glands. If the cancer has spread to the lymph glands there is a high chance that the cancer will come back. To reduce the risk of the cancer recurring, patients are treated with an anticancer drug capecitabine. This study will determine if a simple blood test can predict which patients are at risk for developing side effects from this chemotherapy. In addition, participants of this study will be followed to determine if this same blood test will predict which patients will have their cancer relapse.

DETAILED DESCRIPTION:
Hypothesis:

Recently, the thymidylate synthase gene's promoter has been found to be polymorphic, with variable numbers of tandem repeats of 28 base pairs in length. These polymorphisms have been associated with tumor response to treatment with fluoropyrimidines. The investigators hypothesize that polymorphisms in thymidylate synthase (TS) gene's promoter region are associated with toxicity from capecitabine treatment specifically development of myelosuppression and diarrhea. The investigators hypothesize that a polymorphism in methylene tetrahydrofolate reductase (MTHFR) is also associated with toxicity and efficacy of capecitabine treatment. The investigators speculate that the MTHFR polymorphism only becomes clinically significant by stratifying patients by TS promoter polymorphisms.

Objectives:

1. To determine if polymorphisms in thymidylate synthase's promoter region are associated with development of overall toxicity, diarrhea, neutropenia, or mucositis in patients treated with capecitabine.
2. To determine if a polymorphism in methylene tetrahydrofolate reductase (MTHFR) is associated with development of overall toxicity, diarrhea, neutropenia, or mucositis in patients treated with capecitabine.

Background and Significance:

Capecitabine is a potent antimetabolite that is the currently accepted adjuvant treatment for colorectal cancer. As well, capecitabine is used to treat head and neck cancers, breast cancer and gastric cancer. In 1985, Takeishi et al demonstrated that thymidylate synthase's gene had a satellite in the 5' untranslated region, which consisted of 3 tandem repeats of a 28 base pair sequence. Horie et al demonstrated that these satellites were polymorphic in length due to different numbers of tandem repeats, with 2 length polymorphism existing 2 tandem repeats of 28 base pairs (2R) and 3 tandem repeats of 28 base pairs (3R). Subsequent authors have demonstrated 4 repeats (4R), five repeats (5R) and nine repeats (9R).

Kawakami et al demonstrated that the number of tandem repeats affected TS gene translation. They showed those patients homozygous for 3R alleles had higher TS protein levels and 2R/3R heterozygotes. Using in vitro expression of 2R and 3R genes they demonstrated that the increased protein levels were due to increased translational efficiency of the 3R RNA and not due to increased 3R mRNA expression. These tandem repeats are predictive of response rates of various cancers to fluoropyrimidine cancer chemotherapy. Park et al showed in metastatic colorectal cancer patients treated with capecitabine, the response rate was 14% in patients homozygous for 3R repeats, and 80% in the patients homozygous for 2R repeats. No prospective study has examined if a patient's TS genotype predicts for 5-FU toxicity.

A polymorphism in methylene tetrahydrofolate reductase's (MTHFR) gene may also determine a patient's risk for capecitabine toxicity. A polymorphism in MTHFR exists at position 677, C to T producing a thermolabile and rapidly degraded enzyme. TT homozygotes have increased levels of methylene tetrahydrofolate. Methylene tetrahydrofolate stabilizes binding of 5FU to thymidylate synthase and the complex of TS, 5FU, and methylene tetrahydrofolate is referred to as the ternary complex. I hypothesize that increased stabilization of TS and 5FU due to increased amounts of methylene tetrahydrofolate would lead to increased capecitabine toxicity and efficacy. No study has examined if TT homozygotes have an increased response rate to fluoropyrimidines or increased toxicity.

Dihydropyrimidine dehydrogenase (DPD) deficiency has been identified as the cause of rare severe life threatening reactions to fluoropyrimidines. The first case was reported by Tuchman et al in a 27 year old woman who had undergone adjuvant chemotherapy with cyclophosphamide, methotrexate, and 5-fluoruracil and developed severe neurological complications. Diasio et al reported the second case again in a women being treated with 5-fluoruracil for breast cancer.

A study by Etienne et al has raised questions regarding the utility of DPD activity alone to predict patients at risk for fluoropyrimidine toxicity. They prospectively studied 185 patients treated with 5FU containing chemotherapy regimens. They found a normal distribution of DPD activity with a mean value of 0.222 nmol/min/mg protein. They did not find any correlation between DPD activity and 5FU toxicity.

The investigators propose to study the effect of these two polymorphic enzymes on capecitabine's toxicity in adjuvant colon cancer patients. It is anticipated that patients homozygous for 2R/2R will have higher rates of overall toxicity, diarrhea, neutropenia and mucositis than 3R/3R homozygotes. For MTHFR, we anticipate that TT homozygotes will have higher rates overall toxicity, diarrhea, neutropenia, and mucositis than CC homozygotes. The effect of MTHFR polymorphism on capecitabine's toxicity will be examined controlling for thymidylate synthase genotype.

Methods:

Patients who have been advised to have adjuvant chemotherapy for colorectal cancer will be enrolled. Patients will be treated with standard doses of capecitabine according to the X-ACT study. Toxicities during cycle one will be graded according to National Cancer Institute Common Toxicity Criteria Version 3.0. Dose reductions during cycle one will be recorded.

Investigations:

Prior to starting treatments patients will provide a 10 ml sample of blood which will be used to obtain DNA from white bloods. Patients will be genotyped according to TS and MTHFR genotypes. Plasma will be banked to determined DPD phenotype.

Sample Size Calculation:

The allele frequency of 3R tandem repeats is 0.6 and 2R tandem repeats is 0.417. In 100 patients therefore, I would expect 16 patients with 2R/2R genotypes, 48 with 2R/3R genotypes and 36 with 3R/3R genotypes. It is interesting to note that the incidence of grade 3/4 palmar plantar erythrodysesthesia and diarrhea is on the order of 14 to 16 percent. A sample of 104 patients we would have a power of 0.8 to show a statistically significant difference of 40% between 2R/2R (60%) and 3R/3R (20%).

Statistical Analysis:

Associations between TS genotype and development of grade 1/2 and 3/4 overall toxicity will be examined using the chi square test, with a level of significance of 0.05. Other toxicities of interest, diarrhea, mucositis and neutropenia, will be examined for association with TS genotype chi square test. Similar exploratory analysis will be done for MTHFR phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* High risk Stage II or III colon cancer
* Eastern Cooperative Oncology Group performance status (ECOG P.S.) O or l
* No prior chemotherapy
* Complete tumor resection
* Candidate for and planned to receive standard capecitabine
* Adequate bone marrow reserve

Exclusion Criteria:

* Known DED deficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2005-05; Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada